CLINICAL TRIAL: NCT02523196
Title: Correlation and Comparison of the HepQuant® Disease Severity Index (DSI) With Hepatic Venous Pressure Gradient (HVPG)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-0520; UL1TR001082 (NIH)
Record Dates: First submitted 2015-08-03; First posted 2015-08-14 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Liver Disease
Keywords: Hepatic Venous Pressure Gradient (HVPG) testing; HepQuant-SHUNT; Liver Function
MeSH Terms: conditions — Liver Diseases | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- (HVPG) and HepQuant-SHUNT (HQ-Shunt) (Other): Successful Hepatic Venous Pressure Gradiant (HVPG) testing is required prior to administration of the HepQuant-SHUNT test.
  Comparison of Disease Severity Index (DSI) from HQ-SHUNT with HVPG in identifying patients with cirrhosis and patients with varices.
  Interventions: Drug: HepQuant-SHUNT (Drug and Device) #65,123 (4D-cholate) and IND #65,121 (13C-cholate); Device: Hepatic Venous Pressure Gradient (HVPG)

INTERVENTIONS:
Drug: HepQuant-SHUNT (Drug and Device) #65,123 (4D-cholate) and IND #65,121 (13C-cholate) — The HQ-SHUNT test is being evaluated for safety and effectiveness as an alternative to Hepatic Venous Pressure Gradient (HVPG) testing in patients with liver disease
  Other Names: HQ-SHUNT
Device: Hepatic Venous Pressure Gradient (HVPG) — Hepatic Venous Pressure Gradient (HVPG) is a test for patients with liver disease
  Other Names: (HVPG)

SUMMARY:
This study plans to learn more about a new test to look at liver function, the HepQuant-Shunt (HQ-Shunt). The HQ-Shunt is being evaluated for safety and effectiveness as an alternative to Hepatic Venous Pressure Gradient testing in patients with liver disease.

DETAILED DESCRIPTION:
The goal of this study is to demonstrate the HQ-SHUNT is safe, simple to administer, noninvasive, cost-effective, and well tolerated by patients. This study will compare the HQ-SHUNT to Hepatic Venous Pressure Gradient (HVPG) testing. In this study, 100 consecutive patients with various etiologies of liver disease who have undergone technically successful HVPG testing as standard of care will also undergo HQ-SHUNT testing.

ELIGIBILITY:
Inclusion Criteria:

* Liver disease patient scheduled to have an Hepatic Venous Pressure Gradient (HVPG) procedure
* At time of enrollment, being between the ages of 18 and 75

Exclusion Criteria:

* Concomitant treatment with both a beta blocker and an ACE inhibitor
* Concurrent hepatic malignancy. Patients with a history of treated HCC can be included if there is no evidence of recurrent disease at the time of this study.
* Unstable angina or history of myocardial infarction or congestive heart failure within 6 months prior to enrollment into this study
* Renal insufficiency with chronic kidney disease stage 4 or 5 (GFR < 30 mL/min/1.73m2)
* Crohn's disease or any active intestinal inflammatory condition
* Having had an ileal resection
* Diabetic Gastroparesis
* Pregnancy or intent to become pregnant. Urine pregnancy tests will be performed prior to HQ SHUNT testing.
* Inability to consent for one's self

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Wieland, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver (Leprino Building), Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Everson GT, Shiffman ML, Hoefs JC, Morgan TR, Sterling RK, Wagner DA, Lauriski S, Curto TM, Stoddard A, Wright EC; HALT-C Trial Group. Quantitative liver function tests improve the prediction of clinical outcomes in chronic hepatitis C: results from the Hepatitis C Antiviral Long-term Treatment Against Cirrhosis Trial. Hepatology. 2012 Apr;55(4):1019-29. doi: 10.1002/hep.24752. Epub 2012 Mar 1. PMID 22030902

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects can be excluded if they do not complete the study visit within 60 days of the HVPG testing or if they test positive in a urine pregnancy test the day of the HQ-SHUNT test.
Groups:
- Hepatic Venous Pressure Gradient (HVPG) and HepQuant-SHUNT (HQ: Comparison of Disease Severity Index (DSI) from HQ-SHUNT with HVPG in identifying patients with cirrhosis and patients with varices.
  Successful Hepatic Venous Pressure Gradiant (HVPG) testing is required prior to administration of the HepQuant-SHUNT test.
  Hepatic Venous Pressure Gradient (HVPG): Hepatic Venous Pressure Gradient (HVPG) is a test for patients with liver disease
  HepQuant-SHUNT: The HQ-SHUNT test is being evaluated for safety and effectiveness as an alternative to Hepatic Venous Pressure Gradient (HVPG) testing in patients with liver disease
Period: Overall Study
Arm/Group | Hepatic Venous Pressure Gradient (HVPG) and HepQuant-SHUNT (HQ
Started | 20
Received HVPG | 20
Received HQ Shunt | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HepQuant-SHUNT (HQ-Shunt): Comparison of Disease Severity Index (DSI) from HQ-SHUNT with HVPG in identifying patients with cirrhosis and patients with varices.
  HepQuant-SHUNT: The HQ-SHUNT test is being evaluated for safety and effectiveness as an alternative to Hepatic Venous Pressure Gradient (HVPG) testing in patients with liver disease
Arm/Group | HepQuant-SHUNT (HQ-Shunt)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20
  Non-Wihite | 0
Weight [Mean (Standard Deviation); unit: Kg] | 87.1 (19.7)
Etiology of Liver Disease [Count of Participants; unit: Participants]
  NASH | 9
  HCV | 4
  Autoimmune Hepatitis | 3
  Wilsons Disease | 1
  Budd-Chiari Syndrome | 1
  Cryptogenic | 1
  Other | 1
Fibrosis Stage [Count of Participants; unit: Participants] — Fibrosis stage indicates the severity of scarring of the liver. Possible grades range from F0 to F4, with F0 indicating no scarring and F4 indicating the most severe scarring.
  Participants
    F0 | 2
    F1 | 6
    F2-F3 (F2.5) | 3
    F3 | 3
    F4 | 5
    NA | 1
Steatosis Grade [Count of Participants; unit: Participants]
  Mild, <5% | 4
  Mild, 5 to 33% | 9
  Moderate, 33 to 66% | 4
  Severe, >66% | 1
  NA | 2
Co-Morbid Conditions [Number; unit: participants]
  Obesity | 10
  Diabetes Mellitus | 9
  Hypertension | 8
  Dyslipidemia | 4
  Gout | 1
  Extrahepatic autoimmune disease | 7
  Pulmonary hypertension | 1
  Malignancy | 1
Standard Laboratory Tests: Serum Sodium [Mean (Standard Deviation); unit: mEq/L] | 136 (4)
Standard Laboratory Tests: Creatine, Glucose and Bilirubin [Mean (Standard Deviation); unit: mg/dL]
  Creatine | 0.71 (0.15)
  Glucose | 149 (140)
  Bilirubin | 0.75 (0.34)
Standard Laboratory Tests: AST, Alkaline Phosphatase, ALT [Mean (Standard Deviation); unit: IU/L]
  AST | 46 (36)
  Alkaline Phosphatase | 108 (100)
  ALT | 53 (45)
Standard Laboratory Tests: Albumin [Mean (Standard Deviation); unit: g/L] | 3.79 (.49)
Standard Laboratory Tests: WBC, RBC and Platelets [Mean (Standard Deviation); unit: count/nL]
  WBC | 7.22 (3.06)
  RBC | 4.44 (0.84)
  Platelets | 218.45 (102.56)
Standard Laboratory Tests: Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.38 (2.91)
Standard Laboratory Tests: Hematocrit [Mean (Standard Deviation); unit: %] | 39.60 (7.50)
Standard Laboratory Tests: INR [Mean (Standard Deviation); unit: No units (ratio)] | 1.11 (0.14)
Standard Laboratory Tests: MELD Score [Mean (Standard Deviation); unit: units on a scale] — Model For End-Stage Liver Disease (MELD) scores range from 6 to 40, and is a measure of how severe a patient's liver disease is. Higher scores represent more severe liver disease and a worse outcome.
  units on a scale | 7.35 (1.84)
Standard Laboratory Tests: Child-Turcotte-Pugh (CTP) Score [Mean (Standard Deviation); unit: units on a scale] — The Child-Turcotte-Pugh (CTP) score measures cirrhosis severity. Scores range from 5-15, with higher scores indicating more severe cirrhosis and a worse outcome.
  units on a scale | 5.35 (0.59)

OUTCOME MEASURES:

1. Primary Outcome: Results of HepQuant SHUNT Test: Elimination Rate (IV Phase 1 Only; Min-1)
Description: Compare Disease Severity Index (DSI) from HQ-SHUNT for defining patients with (HVPG ≥6 mmHg) and without (HVPG <6 mmHg) portal hypertension.
Time Frame: Up to 90 minutes
Measure: Mean (Standard Deviation); unit: min-1
Groups:
- HVPG <6 mmHg: Patients without portal hypertension
- HVPG ≥6 mmHg: Patients with portal hypertension
- All Patients: patients with (HVPG ≥6 mmHg) and without (HVPG <6 mmHg) portal hypertension
Arm/Group | HVPG <6 mmHg | HVPG ≥6 mmHg | All Patients
Number analyzed (Participants) | 11 | 9 | 20
min-1 | 0.104 (0.017) | 0.092 (0.023) | 0.099 (0.020)

2. Primary Outcome: Results of HepQuant SHUNT Test: Systemic Clearance
Description: Compare Disease Severity Index (DSI) from HQ-SHUNT for defining patients with (HVPG ≥6 mmHg) and without (HVPG <6 mmHg) portal hypertension. Systemic Clearance (13C-CA; ml min-1)
Time Frame: Up to 90 minutes
Measure: Mean (Standard Deviation); unit: (13C-CA; ml min-1)
Arm/Group | HVPG <6 mmHg | HVPG ≥6 mmHg | All Patients
Number analyzed (Participants) | 11 | 9 | 20
(13C-CA; ml min-1) | 463 (161) | 384 (137) | 427 (152)

3. Primary Outcome: Results of HepQuant SHUNT Test: Apparent Portal Clearance
Description: as for outcome 1
Time Frame: Up to 90 minutes
Measure: Mean (Standard Deviation); unit: d4-CA; ml min-1
Arm/Group | HVPG <6 mmHg | HVPG ≥6 mmHg | All Patients
Number analyzed (Participants) | 11 | 9 | 20
d4-CA; ml min-1 | 1538 (525) | 975 (464) | 1285 (564)

4. Primary Outcome: Results of HepQuant SHUNT Test: Systemic Hepatic Filtration Rate
Description: as for outcome 1
Time Frame: Up to 90 minutes
Measure: Mean (Standard Deviation); unit: ml min-1 kg-1
Arm/Group | HVPG <6 mmHg | HVPG ≥6 mmHg | All Patients
Number analyzed (Participants) | 11 | 9 | 20
ml min-1 kg-1 | 5.30 (1.09) | 4.47 (1.43) | 4.92 (1.29)

5. Primary Outcome: Results of HepQuant SHUNT Test: Portal Hepatic Filtration Rate
Description: as for outcome 1
Time Frame: Up to 90 minutes
Measure: Mean (Standard Deviation); unit: ml min-1 kg-1
Arm/Group | HVPG <6 mmHg | HVPG ≥6 mmHg | All Patients
Number analyzed (Participants) | 11 | 9 | 20
ml min-1 kg-1 | 17.83 (6.37) | 11.11 (5.24) | 14.81 (6.69)

6. Primary Outcome: Results of HepQuant SHUNT Test: SHUNT
Description: Compare Disease Severity Index (DSI) from HQ-SHUNT for defining patients with (HVPG ≥6 mmHg) and without (HVPG <6 mmHg) portal hypertension.
  SHUNT% is The percent of the oral dose of cholate that escapes hepatic extraction
Time Frame: Up to 90 minutes
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | HVPG <6 mmHg | HVPG ≥6 mmHg | All Patients
Number analyzed (Participants) | 11 | 9 | 20
percentage | 29.08 (9.89) | 47.50 (24.24) | 37.37 (19.68)

7. Primary Outcome: Results of HepQuant SHUNT Test: DSI Score
Description: Compare Disease Severity Index (DSI) from HQ-SHUNT for defining patients with (HVPG ≥6 mmHg) and without (HVPG <6 mmHg) portal hypertension.
  DSI range is from 0 to 50. 0 implies no disease; 50 implies severe end-stage disease.
Time Frame: Up to 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale (DSI Score)
Arm/Group | HVPG <6 mmHg | HVPG ≥6 mmHg | All Patients
Number analyzed (Participants) | 11 | 9 | 20
score on a scale (DSI Score) | 14.64 (3.86) | 20.68 (6.30) | 17.36 (5.84)

8. Secondary Outcome: Survey Patients on Their Experience of Having Both HQ-SHUNT and HVPG Procedures.
Description: Overall experience and willingness to repeat 0-10 Scale 0 being no pain, 10 being severe pain 0 being no discomfort, 10 being severe discomfort 0 being no interference with daily life, 10 being unable to carry on activities 0 being very negative experience, 10 being very positive experience 0 being definitely not wanting to have the test again, 10 being very willing to have the test again
Time Frame: Immediately post HepQuant SHUNT test (Baseline up to Day 60)
Population: subjects that underwent HVPG and HQ-Shunt completed surveys
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hepatic Venous Pressure Gradient (HVPG): Successful Hepatic Venous Pressure Gradiant (HVPG) testing is required prior to administration of the HepQuant-SHUNT test.
  Hepatic Venous Pressure Gradient (HVPG): Hepatic Venous Pressure Gradient (HVPG) is a test for patients with liver disease
Arm/Group | Hepatic Venous Pressure Gradient (HVPG) | HepQuant-SHUNT (HQ-Shunt)
Number analyzed (Participants) | 20 | 20
units on a scale
  Pain | 3.9 (3.14) | .35 (.59)
  Discomfort | 4.2 (2.89) | .5 (.89)
  Interfere with Daily Life | 5.9 (3.14) | 1.25 (1.41)
  Overall Experience | 6.2 (2.73) | 9.6 (.68)
  Willingness to Repeat | 5.65 (3.59) | 9.85 (.37)

9. Secondary Outcome: Hours for Test
Description: Number of hours it took for subjects to complete each test
Time Frame: Baseline, up to Day 60
Population: Number of hours
Measure: Number; unit: participants
Arm/Group | Hepatic Venous Pressure Gradient (HVPG) | HepQuant-SHUNT (HQ-Shunt)
Number analyzed (Participants) | 20 | 20
participants
  0-3 hours | 4 | 18
  3-6 hours | 5 | 2
  6-9 hours | 3 | 0
  9-12 hours | 8 | 0

10. Primary Outcome: Results of HepQuant SHUNT Test: STAT
Description: Compare HepQuant STAT test from HQ-SHUNT for defining patients with (HVPG ≥6 mmHg) and without (HVPG <6 mmHg) portal hypertension. HepQuant STAT is a simple "drink and draw" blood-based clearance test that quantifies hepatic impairment from early through late stages of disease.
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: uM/min
Arm/Group | HVPG <6 mmHg | HVPG ≥6 mmHg | All Patients
Number analyzed (Participants) | 11 | 9 | 20
uM/min | 0.61 (0.27) | 1.29 (0.73) | 0.92 (0.62)

ADVERSE EVENTS:
Time Frame: 6 Weeks
Description: no adverse events
Arm/Group | Hepatic Venous Pressure Gradient (HVPG) | HepQuant-SHUNT (HQ-Shunt)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Study did not reach enrollment goal of 110, therefore analysis was limited due to low power

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-08-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT02523196/Prot_SAP_001.pdf
  • Informed Consent Form (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT02523196/ICF_000.pdf